CLINICAL TRIAL: NCT00410007
Title: The Effect of High and Low Sodium Intake on Urinary Aquaporin-2 in Autosomal Dominant Polycystic Kidney Disease, During Basal Conditions and After Hypertonic Saline Infusion.
Brief Title: The Effect of High and Low Sodium Intake on Urinary Aquaporin-2 in Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Cannillo (Other)
Responsible Party: Sponsor-Investigator, Carolina Cannillo, Principal Investigator, PhD, MD, Regional Hospital Holstebro
Organization: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: med.res.hos.2006.cc.03
Record Dates: First submitted 2006-12-10; First posted 2006-12-12 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Polycystic Kidney, Autosomal Dominant
Keywords: ADPKD; Urinary Aquaporin-2; ENaC; Fractional sodium excretion; High/low sodium diet
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Patients with ADPKD, HS (Other): Each subject was studied on 2 separate days at least 3 weeks apart. During 4 days before the study day, the subjects consumed either a high sodium diet or a low sodium diet in randomized order (HS-LS/ LS-HS). On the study day a hypertonic saline infusion was given.
  Interventions: Behavioral: High Sodium Diet; Behavioral: Hypertonic saline infusion
- Patients with ADPKD, LS (Other): Each subject was studied on 2 separate days at least 3 weeks apart. During 4 days before the study day, the subjects consumed either a high sodium diet or a low sodium diet in randomized order (HS-LS/ LS-HS). On the study day a hypertonic saline infusion was given.
  Interventions: Behavioral: Low Sodium Diet; Behavioral: Hypertonic saline infusion
- Healthy Control Subjects, HS (Other): Each subject was studied on 2 separate days at least 3 weeks apart. During 4 days before the study day, the subjects consumed either a high sodium diet or a low sodium diet in randomized order (HS-LS/ LS-HS). On the study day a hypertonic saline infusion was given.
  Interventions: Behavioral: High Sodium Diet; Behavioral: Hypertonic saline infusion
- Healthy Control Subjects, LS (Other): Each subject was studied on 2 separate days at least 3 weeks apart. During 4 days before the study day, the subjects consumed either a high sodium diet or a low sodium diet in randomized order (HS-LS/ LS-HS). On the study day a hypertonic saline infusion was given.
  Interventions: Behavioral: Low Sodium Diet; Behavioral: Hypertonic saline infusion

INTERVENTIONS:
Behavioral: High Sodium Diet — 250-350 mmol
  Arms: Healthy Control Subjects, HS; Patients with ADPKD, HS
Behavioral: Low Sodium Diet — 25-35 mmol
  Arms: Healthy Control Subjects, LS; Patients with ADPKD, LS
Behavioral: Hypertonic saline infusion — 7 ml/ kg of 3% saline were given over 30 minutes.

SUMMARY:
The aim of the study is to test the following hypotheses:

1. that the function and/or regulation of AQP2 and /or ENaC in the principal cells is abnormal in autosomal dominant polycystic kidney disease.
2. if an abnormal function of the principal cells is present in autosomal dominant polycystic kidney disease, this will become more pronounced at high and low sodium intake.

DETAILED DESCRIPTION:
Recruitment:

The patients with ADPKD are recruited from the Outpatient Nephrology Clinic of the Department of Medicine, Holstebro Hospital (Holstebro, Denmark). The control subjects are recruited by advertising in public institutions and private companies.

Number of Subjects:

A difference in u-AQP2CR of 40 ng/mmol is considered the minimal relevant difference. A sample size of 10 subjects, who can be evaluated, has 80% power to detect this difference assuming a level of signiﬁcance of 5% and an SD of 30 ng/mmol. Because a few subjects are expected to drop out, 14-15 subjects will be included in each group.

Experimental Procedure Before the Study Day:

Five days before the study day, the subjects collect a standardized, HS (300 mmol sodium/day/17.5 g salt/day) or LS (30 mmol sodium/day/1.8 g salt/day), 4-day diet from the hospital kitchen. Depending on the individually estimated energy requirement, the participants are given either a diet of 8,000 or 11,000 kJ/day. The energy distribution is 55% carbohydrates, 15% proteins, and 30% lipids. The 4-day diet is started the following morning. The ﬂuid intake is also standardized during the 4 days. The subjects are asked to drink exactly 250 ml/1,000 kJ/day and to abstain from coffee, tea, and alcoholic beverages. The subjects are instructed to keep their physical activity unchanged during the two experiments and to abstain from hard training. The subjects have to collect their urine for 24 h the day before the study day.

Experimental Procedure on the Study Day:

On the study day, the subjects are asked to drink 175 ml of water every 30 min from 7:00 AM. The subjects arrive at the department at 8:00 AM. Peripheral iv lines are inserted into the antecubital veins of both forearms, one for infusion of 51Cr-EDTA and hypertonic saline, and one for withdrawal of blood samples. The subjects will be kept in the supine position from 8:00 AM to 1:30 PM except during voiding, which will take place in the sitting or standing position. At 8:30 AM, a priming dose of 51Cr-EDTA is administered, followed by sustained infusion. After 60 min of equilibration, the study will continue with ﬁve clearance periods, the ﬁrst two of 30-min duration (P1-P2), the last three of 60-min duration (P3-P5). The ﬁrst two clearance periods are baseline periods. At 10:30 AM, 7 ml/kg of 3% saline is given over 30 min. Blood pressure and heart rate are measured every 30 min from 9:30 AM to 1:30 PM. Urine is collected in each clearance period and analyzed for sodium, osmolality, u-AQP2, u-ENaC-betaCR, u-cAMP, u-PGE2, and 51CrEDTA. Blood samples will be drawn every 30 min from 9:30 AM to 10:30 AM and every hour from 11:30 AM to 1:30 PM, and will be analyzed for sodium, osmolality, and 51Cr-EDTA. In addition, analysis of p-AVP, p-Renin, p-ANG II, p-Aldo, p-ANP, and p-BNP will be performed from blood samples drawn at 10:30 AM, 11:30 AM, 12:30 PM, and 1:30 PM.

Statistics:

Statistical analyses will be performed using SPSS version 15 (SPSS, Chicago, IL). Single baseline values are obtained by taking the weighted average of the measurements from the two baseline periods. The baseline values of the two groups will be compared by Student's t-test. The baseline values during HS and LS intake will be compared by paired samples t-tests. The investigators will use the "General Linear Model Repeated Measures" procedure in SPSS with time as the within-subject factor and group as the between-subject factor to compare the effect variables in patients and controls. The changes in response to the hypertonic saline infusion in each group will be analyzed with the General Linear Model Repeated Measures procedure with time as the within-subject factor and paired samples t-tests with Bonferroni correction as post hoc tests. P values Recruitment The patients with ADPKD will be recruited from the Outpatient Nephrology Clinic of the Department of Medicine, Holstebro Hospital (Holstebro, Denmark). The control subjects will be recruited by advertising in public institutions and private companies.

Number of Subjects A difference in u-AQP2CR of 40 ng/mmol is considered the minimal relevant difference. A sample size of 10 subjects, who could be evaluated, has 80% power to detect this difference assuming a level of signiﬁcance of 5% and an SD of 30 ng/mmol. Because a few subjects are expected to drop out, 14-15 subjects will be included in each group.

Experimental Procedure Before the Study Day Five days before the study day, the subjects will collect a standardized, HS (300 mmol sodium/day/17.5 g salt/day) or LS (30 mmol sodium/day/1.8 g salt/day), 4-day diet from the hospital kitchen. Depending on the individually estimated energy requirement, the participants will be given either a diet of 8,000 or 11,000 kJ/day. The energy distribution will be 55% carbohydrates, 15% proteins, and 30% lipids. The 4-day diet will start the following morning. The ﬂuid intake is also standardized during the 4 days. The subjects are asked to drink exactly 250 ml/1,000 kJ/day and to abstain from coffee, tea, and alcoholic beverages. The subjects will be instructed to keep their physical activity unchanged during the two experiments and to abstain from hard training. The subjects have to collect their urine for 24 h the day before the study day.

Experimental Procedure on the Study Day On the study day, the subjects are asked to drink 175 ml of water every 30 min from 7:00 AM. The subjects arrive at the department at 8:00 AM. Peripheral iv lines will be inserted into the antecubital veins of both forearms, one for infusion of 51Cr-EDTA and hypertonic saline, and one for withdrawal of blood samples. The subjects will be kept in the supine position from 8:00 AM to 1:30 PM except during voiding, which will take place in the sitting or standing position. At 8:30 AM, a priming dose of 51Cr-EDTA is administered, followed by sustained infusion. After 60 min of equilibration, the study will continue with ﬁve clearance periods, the ﬁrst two of 30-min duration (P1-P2), the last three of 60-min duration (P3-P5). The ﬁrst two clearance periods are baseline periods. At 10:30 AM, 7 ml/kg of 3% saline is given over 30 min. Blood pressure and heart rate will be measured every 30 min from 9:30 AM to 1:30 PM. Urine is collected in each clearance period and analyzed for sodium, osmolality, u-AQP2, u-ENaC-betaCR, u-cAMP, u-PGE2, and 51CrEDTA. Blood samples will be drawn every 30 min from 9:30 AM to 10:30 AM and every hour from 11:30 AM to 1:30 PM, and will be analyzed for sodium, osmolality, and 51Cr-EDTA. In addition, analysis of p-AVP, p-Renin, p-ANG II, p-Aldo, p-ANP, and p-BNP will be performed from blood samples drawn at 10:30 AM, 11:30 AM, 12:30 PM, and 1:30 PM.

Statistics Statistical analyses will be performed using SPSS version 15 (SPSS, Chicago, IL). Single baseline values are obtained by taking the weighted average of the measurements from the two baseline periods. The baseline values of the two groups will be compared by Student's t-test. The baseline values during HS and LS intake will be compared by paired samples t-tests. The investigators will use the "General Linear Model Repeated Measures" procedure in SPSS with time as the within-subject factor and group as the between-subject factor to compare the effect variables in patients and controls. The changes in response to the hypertonic saline infusion in each group will be analyzed with the General Linear Model Repeated Measures procedure with time as the within-subject factor and paired samples t-tests with Bonferroni correction as post hoc tests. P values ≤0.05 will be considered signiﬁcant.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women
* age 18-65 years
* BMI between 18,5-30,0 kg/m2
* ADPKD, diagnosed by the following findings on ultra scan:

  * for patients without ADPKD family history: > 5 bilateral cysts
  * for patients with ADPKD family history: < 30 years: 2 cysts (unilateral or bilateral) 30-60 years: 2 or more bilateral cysts > 60 years: 4 or more bilateral cysts
* Kidney function: stadium 1-4.

Exclusion Criteria:

* Other kidney disease
* Anamnestic or clinical signs of acute myocardial infarction, atrial fibrillation, heart valve disease or chronic heart failure
* Anamnestic or clinical signs of disease in lungs, liver,endocrine organs or brain or neoplastic disease
* Family history of rupture of intracerebral aneurisms
* Alcohol or drug abuse
* Smoking
* Medical treatment arat form antihypertensives and oral anticonceptives
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-10; Primary Completion 2010-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
u-AQP-2CR | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  Urinary Aquaporin-2 corrected for creatinine

SECONDARY OUTCOMES:
u-ENaC (beta)CR | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  Urinary ENaC (beta) corrected for creatinine
FENa | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  fractional sodium excretion
CH2O | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  Free water excretion
u-cAMP | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  urinary excretion of cAMP
uPGE-2 | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  urinary excretion of PGE-2
GFR | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  glomerular filtration rate
p-vasopressin | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  plasma concentration of vasopressin
p-aldosterone. | Before and after hypertonic saline infusion after 4 days on high and low sodium diet, respectively.
  plasma concentration of aldosterone

CONTACTS AND LOCATIONS:
Overall Officials: Erling B. Pedersen, Professor, Study Chair — Department of Medical Research, Holstebro Hospital, Denmark; Carolina C. Graffe, MD, Principal Investigator — Department of Medical Research, Holstebro Hospital, Denmark
Locations (1):
- Department of Medical Research, Holstebro Hospital, Holstebro, Denmark